CLINICAL TRIAL: NCT00078715
Title: An Investigation of a Pharmacologic Strategy to Bring About Rapid (Next Day) Antidepressant Effects
Brief Title: Rapid Antidepressant Effects of Yohimbine in Major Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Carlos Zarate, M.D., Chief of Experimental Therapeutics and Pathophysiology Branch of NIMH, DIRP, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 040091; 04-M-0091 (Other: CNS-IRB, NIH)
Record Dates: First submitted 2004-03-04; First posted 2004-03-05 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Depression, Involutional; Major Depresssion
Keywords: Yohimbine; Sleep Deprivation; Depression; Mood Disorder; Fast; Affective Disorder; Rapid Onset; Major Depression; MDD
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Deprivation; Depression; Mood Disorders; Fasting | interventions — Yohimbine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yohimbine then Placebo (Experimental): Participants are randomized to receive yohimbine 0.125 mg/kg administered over 3 minutes during REM sleep. After 8 days they receive placebo administered over 3 minutes during REM sleep.
  Interventions: Drug: Yohimbine hydrochloride; Drug: Placebo
- Placebo then Yohimbine (Experimental): Participants are randomized to receive placebo administered over 3 minutes during REM sleep. After 8 days they receive yohimbine 0.125 mg/kg administered over 3 minutes during REM sleep.
  Interventions: Drug: Yohimbine hydrochloride; Drug: Placebo

INTERVENTIONS:
Drug: Yohimbine hydrochloride — Participants receive yohimbine 0.125 mg/kg administered over 3 minutes during REM sleep.
Drug: Placebo — Participants receive an inactive equivalent of yohimbine 0.125 mg/kg administered over 3 minutes during REM sleep.

SUMMARY:
This study examines if Yohimbine, when given during the sleep cycle, will improve symptoms of depression within a matter of hours.

Purpose: This study will examine whether the drug yohimbine, given at a specific time during the sleep cycle, produces chemical changes in the brain similar to those that occur with sleep deprivation. It will also see if yohimbine can induce rapid (next day) antidepressant effects in patients with major depression. Total sleep deprivation for 36 hours improves mood in most patients with major depression in a matter of hours, but the response is usually short-lived. Understanding the chemical changes that occur in the body during sleep deprivation may help in the development of a rapidly acting antidepressant.Patients with major depressive disorder between 18 and 65 years of age may be eligible for this study. Candidates are screened with a medical and psychiatric history, physical examination, electrocardiogram, and blood and urine tests. Participants are hospitalized at the NIH Clinical Center for the study, as follows: Drug-free period: Patients are tapered off their anti-depression medications and remain drug-free for 1 week before beginning study phase 1. Study phase 1: Patients undergo sleep deprivation for 36 hours. Those whose depression improves with sleep deprivation initially and then worsens continue to phase 2. The day after sleep deprivation, patients undergo a lumbar puncture (spinal tap). For this test, a local anesthetic is given and a needle is inserted in the space between the bones in the lower back where the cerebrospinal fluid circulates below the spinal cord. A small amount of fluid is collected through the needle. Study phase 2: Patients spend 1 night in the sleep lab. A catheter (plastic tube) is placed in a vein in each arm-one to give yohimbine and the other to draw blood samples. A small monitor cuff is placed on a finger to measure the patient's blood pressure and blood oxygen levels during the night. While asleep, the patient receives a dose of yohimbine or placebo, given over 3 minutes. A lumbar puncture is done the following morning. Patients receive no medications for 6 days, and then the sleep lab procedure is repeated. Patients who received yohimbine in the previous experiment are switched to placebo, and those who were given placebo are switched to yohimbine.

DETAILED DESCRIPTION:
Sleep deprivation is one of the only interventions that have consistently been demonstrated to produce rapid antidepressant effects. The mechanisms by which sleep deprivation brings about rapid antidepressant effects remain to be elucidated. It is noteworthy, however, that recent genomic and proteomic studies have shown that acute sleep deprivation rapidly brings about an upregulation of several mediators of neuronal plasticity, most notably CREB and BDNF. Intriguingly, these are the very same molecules that are upregulated by chronic antidepressants, and are believed to underlie the delayed therapeutic effects of most antidepressants. Additional investigation of the regulation of CREB and BDNF by sleep deprivation has revealed that these changes are critically dependent upon the activation of the noradrenergic system. This is particularly noteworthy, since the locus coeruleus (LC) noradrenergic projection is quiescent only during rapid eye movement sleep (REM), when the target tissues display their greatest sensitivity; indeed, the temporal dissociation between the firing of the LC noradrenergic neurons, and the sensitivity of its postsynaptic targets in the cortex may have considerable relevance for the antidepressant effects of sleep deprivation. In this context, biological rhythms have the capacity to temporally dissociate biochemical processes, and imposing a temporal coincidence on normally dissociated events can have striking and unexpected effects. Thus, it is our hypothesis that activating the normally quiescent noradrenergic system during REM sleep (i.e. when its postsynaptic target system displays its greatest sensitivity) will robustly upregulate CREB and BDNF, thereby bringing about a rapid antidepressant effect. We propose to activate the noradrenergic system during REM sleep by infusing an alpha(2) antagonist, yohimbine. Since it is our hypothesis that activating the noradrenergic system during REM sleep will bring about an antidepressant effect by a similar mechanism as sleep deprivation, we will "enrich" our sample with sleep deprivation responders in this pilot study.

Patients, ages 18 to 65 with a diagnosis of major depressive disorder, currently depressed without psychotic features will be recruited into this study. This experimental proof-of-concept study has two Study Phases. Study Phase I consists of total sleep deprivation. Responders to total sleep deprivation who subsequently relapse will enter Study Phase II. Study Phase II is a double-blind crossover administration of either intravenous yohimbine or saline solution during REM sleep.

The specific aim of this study is to assess the efficacy of a single dose of intravenous yohimbine hydrochloride (0.125 mg/kg given over 3 minutes) compared with placebo in improving overall depressive symptomatology when administered during REM sleep.

Our primary hypothesis is that the intravenous use of an alpha(2) antagonist in patients with major depression during REM sleep will activate the LC and thus increase noradrenergic activity during a time when the LC is normally quiescent- namely REM sleep. If the hypothesis that it is the timing of the activation of the noradrenergic system that is crucial in the antidepressant effect of sleep deprivation is correct then an acute antidepressant effect should be observed in patients despite minimal to no disruption of sleep.

Assuming that 10% will drop out of the study, then a minimum of 25 patients is necessary in order to obtain a minimum of 8 patients with major depression who will complete the double-blind crossover phase of the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Male or female subjects, 18 to 65 years of age.

Female subjects of childbearing potential must be using a medically accepted means of contraception.

Each subject must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.

Subjects must fulfill DSM-IV criteria for Major Depression, based on clinical assessment and confirmed by a structured diagnostic interview, SCID-P.

Subjects must have an initial score of at least 18 on the 21-item HDRS at screen and at baseline of TSD and Study Phase II.

Subjects with a greater than 25% decrease in the 21-item HDRS total scores between screen and baseline of TSD will be dropped from the study.

EXCLUSION CRITERIA:

Subjects with documented uncontrolled hypertension in the 30 days prior to Study Period I, or have a systolic blood pressure greater than or equal to 140 and/or diastolic blood pressure greater than or equal to 90 on 3 or more readings during the drug-free period.

Apnea/hypopnea index is greater than 15 episodes per minute.

Presence of psychotic features or a diagnosis of Schizophrenia or any other psychotic disorder as defined in the DSM-IV.

Subjects with current DSM-IV diagnosis of generalized anxiety disorder, panic disorder, or posttraumatic stress disorder.

Subjects with a history of DSM-IV drug or alcohol dependency or abuse (including for nicotine) within the preceding 3 months.

Female subjects who are either pregnant or nursing.

Serious, unstable illnesses including hepatic, renal gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.

DSM-IV diagnosis of primary sleep disorder.

Subjects with uncorrected hypothyroidism or hyperthyroidism.

Subjects with one or more seizures without a clear and resolved etiology.

Documented history of hypersensitivity or intolerance to yohimbine.

Treatment with a reversible MAOI within 4 weeks prior to Study Phase II.

Treatment with fluoxetine within 3 weeks prior to Study Phase II.

Treatment with any other concomitant medication not allowed 7 days prior to Study Phase II.

Treatment with clozapine or ECT within 3 months prior to Study Phase I.

Judged clinically to be at serious suicide risk.

Previous nonresponse to total sleep deprivation treatment.

STUDY PHASE II:

INCLUSION CRITERIA

Same as above plus:

Response to total sleep deprivation (40% decrease in the HAM-D6) followed by:

Depressive relapse (score of at least 18 on the 21-item HDRS and no longer meets response criteria) prior to Study Period II.

EXCLUSION CRITERIA:

YMRS total score of greater than or equal to 12 within 24 hours of yohimbine administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2004-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — Experimental Therapeutics and Pathophysiology Branch, DIRP, NIMH
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Duman RS. Synaptic plasticity and mood disorders. Mol Psychiatry. 2002;7 Suppl 1:S29-34. doi: 10.1038/sj.mp.4001016. PMID 11986993
- [Background] Poo MM. Neurotrophins as synaptic modulators. Nat Rev Neurosci. 2001 Jan;2(1):24-32. doi: 10.1038/35049004. PMID 11253356
- [Background] Cirelli C, Tononi G. Differential expression of plasticity-related genes in waking and sleep and their regulation by the noradrenergic system. J Neurosci. 2000 Dec 15;20(24):9187-94. doi: 10.1523/JNEUROSCI.20-24-09187.2000. PMID 11124996
- [Derived] Ibrahim L, Duncan W, Luckenbaugh DA, Yuan P, Machado-Vieira R, Zarate CA Jr. Rapid antidepressant changes with sleep deprivation in major depressive disorder are associated with changes in vascular endothelial growth factor (VEGF): a pilot study. Brain Res Bull. 2011 Aug 10;86(1-2):129-33. doi: 10.1016/j.brainresbull.2011.06.003. Epub 2011 Jun 16. PMID 21704134

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with major depression were recruited to participate in the study at the Clinical Center on the main campus of the National Institutes of Health in Bethesda, Maryland. Recruiting began in 2004.
Pre-assignment Details: 11 participants were run through a sleep deprivation procedure and 6 of those had a significant improvement in depression. These 6 sleep deprivation responders were randomized in the crossover yohimbine study.
Groups:
- Placebo Then Yohimbine: Participants are randomized to blindly receive placebo for 8 days then yohimbine for the same.
- Yohimbine Then Placebo: Participants are randomized to blindly receive yohimbine for 8 days then placebo for the same.
Period: First Intervention
Arm/Group | Placebo Then Yohimbine | Yohimbine Then Placebo
Started | 2 | 4
Completed | 2 | 4
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo Then Yohimbine | Yohimbine Then Placebo
Started | 2 | 4
Completed | 2 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.17 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (6 Items)
Description: The 6 item Hamilton Depression Rating Scale is a measurement of the severity of depression with a range of scores from 0 to 24, where 24 indicates the most severe depression.
Time Frame: Once per day, where the primary comparison involves an average over the full study after controlling for baseline
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- Placebo: Participants are randomized to blindly receive placebo for 8 days.
- Yohimbine: Participants are randomized to blindly receive yohimbine for 8 days.
Arm/Group | Placebo | Yohimbine
Number analyzed (Participants) | 6 | 6
Units on a scale | 8.776 (1.141) | 9.780 (1.141)
Statistical Analysis 1: Comparison: Placebo vs Yohimbine; The hypothesis was that yohimbine would provide lower levels of depression than placebo. Initial estimates of sample size assumed a minimum of 25 patients were required to detect differences in depression; Test type: Superiority or Other; p = .527, Mixed Models Analysis — The significance level reflects the direct comparison of drugs after factoring out baseline depression levels; A linear mixed model was used with factors for drug, time of evaluation, the drug by time interaction, and a baseline depression covariate; Mean Difference (Net) = -1.004, 95% CI 2-sided [-4.260 to 2.251], Standard Error of Mean 1.141

ADVERSE EVENTS:
Arm/Group | Placebo | Yohimbine
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Yohimbine (N=6)
Difficulty sleeping (Nervous system disorders) | 0 (0) | 2 (2)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Taste abnormality (General disorders) | 0 (0) | 1 (1)
Increased urination (Renal and urinary disorders) | 0 (0) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sweating (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No